CLINICAL TRIAL: NCT00078455
Title: A Phase II Study of ILX651 Administered Intravenously Daily for Five Consecutive Days Once Every 3 Weeks in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Carcinoma
Brief Title: Study of ILX651 in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILX651-231
Record Dates: First submitted 2004-02-25; First posted 2004-03-01 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Non-Small-Cell Lung Carcinoma
Keywords: NSCLC; Non-small Cell Lung Cancer; Non-small Cell Lung Carcinoma; Locally Advanced NSCLC; Metastatic NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tasidotin

INTERVENTIONS:
Drug: ILX651

SUMMARY:
This is a Phase II, non-randomized, open label study of ILX651 in patients with locally advanced or metastatic non-small cell lung carcinoma (NSCLC). Approximately 60 patients will be enrolled in this study that is expected to last 18 months. All patients will be treated with ILX651 administered intravenously (IV) daily for 5 consecutive days once every 21 days. The primary objective of this study is to determine the overall response rate. The secondary objectives are to determine the progression free survival, duration of response, time to tumor progression, survival, safety/tolerability of ILX651, and to evaluate pharmacokinetic profile.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced or metastatic NSCLC previously treated with 2 prior chemotherapy regimens (not including prior adjuvant therapy for stage I or II disease).
* Disease recurrence or progression after prior therapy with a platinum-based and a taxane-based regimen, given either concurrently or separately.
* Measurable disease. Measurable lesions should be outside the field of radiation. Where measurable lesions are within a previously irradiated field, there must be objective evidence of progression of the lesion prior to patient enrollment.
* Male or female patients greater than or equal to 18 years of age.
* ECOG performance status of 0 or 1.
* Must have adequate organ and immune system function as indicated by the following laboratory values, obtained less than or equal to 2 weeks prior to registration: A. Absolute neutrophil count (ANC) greater than or equal to 1.5 x 1,000,000,000. B. Hemoglobin greater than or equal to 9.0 g/dL. C. Platelet count greater than or equal to 100 x 1,000,000,000/L. D. Serum creatinine or calculated creatinine clearance less than or equal to 1.5 mg/dL or greater than or equal to 60 mL/min. E. Serum total bilirubin within limits of normal values. F. AST and ALT less than or equal to 2 times the upper limit of normal (ULN). G. Alkaline phosphatase within limits of normal values
* Anti-cancer therapy, major surgery, or irradiation must have been completed at least 3 weeks before enrollment in this study. Patient must have recovered from the acute side effects incurred as a result of previous therapy.
* Female patients with childbearing potential must have a negative pregnancy test within 7 days of study enrollment. Men and women of reproductive potential must use an effective contraceptive method while enrolled in the study.
* Signed informed consent (includes HIPAA authorization).

Exclusion Criteria:

* Patients with uncontrolled congestive heart failure or angina, patients with a history of myocardial infarction within 2 months of enrollment, or patients with cardiac functional capacity Class III or IV as defined by the New York Heart Association Classification.
* Previously treated with > 2 prior chemotherapy regimens for advanced or metastatic disease.
* Prior radiotherapy to the only site of measurable disease.
* Known hypersensitivity to study drug or its analogs.
* Use of investigational agents within previous 30 days.
* Known, active infection, or known HIV positive or presence of an AIDS related illness.
* Active secondary malignancy except minor skin cancers.
* Presence of symptomatic active brain metastases, including leptomeningeal involvement.
* Any significant concurrent disease or illness, or psychiatric disorders or alcohol or chemical abuse that would, in the opinion of the investigator, compromise patient safety or compliance, or interfere with the interpretation of study results.
* Pregnant or lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-12; Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - US Oncology/ Arizona Clinical Research Center, Tucson, Arizona
  - Cancer Institute Medical Group, Santa Monica, California
  - Anshutz Cancer Pavillion, Aurora, Colorado
  - US Oncology / Ocala Oncology, Ocala, Florida
  - US Oncology / Central Indiana Cancer Centers, Indianapolis, Indiana
  - Hematology and Oncology Specialists, New Orleans, Louisiana
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - US Oncology / Texas Cancer Center, Dallas, Texas
  - Joe Arrington Cancer Center, Lubbock, Texas
  - US Oncology / Tyler Cancer Center, Tyler, Texas